CLINICAL TRIAL: NCT04661241
Title: MRI-guided Personalized Targeting of the Ventral Intermediate Nucleus (VIM)/Dentato-rubro-thalamic Tract (DRT) for the MRgFUS Tremor Treatment
Brief Title: Mapping the Target for the MRgFUS Treatment of Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 20-00981
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Tremor, Essential; Parkinson's Disease
Keywords: Tremor; Parkinson's Disease; MRgFUS; magnetic resonance-guided focused ultrasound
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Tremor

STUDY DESIGN:
Intervention Model Description: All patients in this study will be recruited from New York University Langone Health in cooperation with the NYU Neurosurgery and the Center for Neuromodulation. The Department of Neurosurgery will make initial contact with prospective patients who will undergo the MRgFUS tremor treatment. The patient's treating physician will determine suitability based on the subject's known clinical status and ability to be informed consent to participate in the study.
Who Masked: Care Provider
Masking Description: As a pilot study, the results of our method will be blinded to the clinician who will operate the MRgFUS tremor therapy in order to compare the locations of the proposed target, surgical lesion and stereotactic coordinates.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Scan (Experimental): The proposed sequence (<15 minutes) will be added as a supplementary sequence only for the preoperative imaging if subjects agree to participate.
  Interventions: Other: Automatic DRT/VIM target-recognition method using MR-SISET and ML approaches
- Current Clinical Practice (Active Comparator): All patients will undergo a routine clinical preoperative MRI of the brain under general anesthesia to reduce movement artifacts.
  Interventions: Other: Routine clinical MRI protocol

INTERVENTIONS:
Other: Automatic DRT/VIM target-recognition method using MR-SISET and ML approaches — The proposed sequence (<15 minutes) will be added as a supplementary sequence only for the preoperative imaging for subjects who agree to participate: a 3D multi-echo GRE sequence will be performed during a preoperative MR imaging, using the following parameters: field of view = 220x170x75 mm3, matrix = 176x136x60, 1.25-mm isotropic resolution, flip angle = 22 degrees, TR = 92 ms, 20 TEs = 1.90 - 45.98 ms with echo spacing of 2.32 ms, bandwidth = 840 Hz/pixel.
  Arms: Investigational Scan
Other: Routine clinical MRI protocol — MRI will be performed using 3T scanner (Skyra, Siemens, Erlangen, Germany). All patients will undergo preoperative MRI of the brain including routine clinical MRI protocol (T1-/T2-weighted and diffusion imaging) under general anesthesia to reduce movement artifacts.
  Arms: Current Clinical Practice

SUMMARY:
The purpose of this investigation is to determine the optimal DRT/VIM target location and its safety margins based on MR-SISET imaging features by comparing with postoperative lesions and clinical outcomes in patients with tremor who will undergo the MRgFUS tremor therapy.

DETAILED DESCRIPTION:
Magnetic susceptibility is an important source of contrast in MRI, which arises from the subtle field perturbations generated by inter-molecular interaction in response to an external magnetic field. The DRT tract consists mainly of axon fibers covered by myelin sheaths that cause magnetic susceptibility variations. In addition, magnetic susceptibility of fiber bundle is in fact anisotropic. Such distinctive features of the DRT can generate a unique type of susceptibility contrast with respect to its neighboring thalamic tissues, yet clinically practical protocols are lacking. This study will utilize a novel MR susceptibility-based method, termed 'MR Susceptibility Imaging with Short Echo Time (MR-SISET)' which leverages short echo times to realize high contrast for direct and individualized DRT targeting. Combined with machine learning (ML) approaches, an automatic, operator-independent DRT-recognition will be achieved. This could provide a valid support to operators in the surgical planning and significantly improve the current operative methodology.

MR imaging will be done on a 3T MRI Magnet at the NYU Langone Health. All patients will undergo a routine clinical preoperative MRI of the brain under general anesthesia to reduce movement artifacts. The proposed sequence (<15 minutes) will be added as a supplementary sequence only for the preoperative imaging for subjects who agree to participate. The operator/clinician will be blinded to the results of this study for the MRgFUS treatment. A routine clinical postoperative MRI will be performed prior to discharge by the clinician, typically the following day of the MRgFUS treatment. The severity of tremor will be assessed before and after the treatment (~6 weeks). Postoperative clinical data will be retrieved to get a surgical target lesion and clinical outcome after treatment in order to confirm our method.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Any ethnic background
* History of a primary diagnosis of essential tremor or Parkinson's disease
* Present for the MRgFUS tremor treatment
* Ability to understand and agree to informed consent as determined by referring physician

Exclusion Criteria:

* Inability to give informed consent
* Contraindications for MRI, including

  1. Intracranial clips
  2. Metal implants
  3. External metallic devices/objects/clips within 10 mm of the head
  4. Suspected or confirmed metal in eyes (history of welding or similar activity)
  5. Cardiac pacemaker
  6. Pregnant or potentially pregnant - pregnancy tests will be offered to women of childbearing age at no cost to the patient. (A SOC pregnancy test (Urine test) will be done for women of child bearing age if requested/required at the time of check-in at Tisch.This will be billed to the research study). The result of the test (if performed) will be added to the patient's chart in EPIC.
  7. No vulnerable populations will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Tremor improvement | 6 weeks
  A routine clinical follow-up will be performed to assess the severity of tremor after the treatment (~ 6 weeks) by the clinician. Patients will be categorized into three groups based on their outcome: a good clinical outcome (>65% tremor improvement), a moderate outcome (>33%, but <66% tremor improvement) and a poor outcome (<33% tremor improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Sohae Chung, MD, Principal Investigator — NYU Langone; Timothy Shepherd, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to sohae.chung@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to sohae.chung@nyulangone.org.